CLINICAL TRIAL: NCT01772511
Title: BrUOG 274: Do Patients Participating In Oncology Clinical Trials Understand the Informed Consent Form?
Brief Title: Do Patients Participating In Oncology Clinical Trials Understand the Informed Consent Form?
Status: Completed | Type: Observational
Sponsor: Andrew Sch umacher (Other)
Responsible Party: Sponsor-Investigator, Andrew Sch umacher, Principal Investigator, Brown University
Organization: Brown University (Other)
Other Study IDs: 274
Record Dates: First submitted 2013-01-14; First posted 2013-01-21 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2014-12

CONDITIONS: Cancer; Oncology Problem
Keywords: questionnaire; prior therapy; prior study volunteer; prior study patient; cancer; oncology
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Questionnaire: Patients will be asked by a member of the research team if they would like to participate in this study evaluating patients' comprehension of the informed consent for the oncology treatment study that they are participating in. Patients will be consented and will be told that, at their next clinical visit, they will be given the questionnaire to complete. They will be given the option to complete the questionnaire on site after being given the document or have the ability to mail the completed questionnaire into the research office once completed. If the questionnaire is not returned within 2-weeks, the participant will be approached again during their normal clinical visit and asked if they still wish to participate in this study.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — All patients entering on this trial will have been enrolled on an oncology clinical trial and are receiving active anti-cancer treatment on that study.

SUMMARY:
The purpose of this study is to assess patients' understanding of clinical trials and to help researchers understand which areas of the informed consent need better explanation for future cancer clinical trial patients.

DETAILED DESCRIPTION:
Obtaining informed consent as part of a clinical study is a cornerstone of current day medical ethics; however, this has not always been the case. The development of the informed consent has been necessitated out of abuses committed in the name of medicine.

Informed consents have become increasing lengthy and complex. It is not unusual for an Oncology Clinical Research informed consent to be greater than 20 pages. Investigators will utilize the QuIC-A survey to evaluate patient understanding of the basic elements of informed consent required by federal regulations. The QuIC-A survey has been condensed from 20 questions to 14 questions by eliminating the 6 phase specific questions. The remaining 14 questions are designed irrespective of phase and address the basic elements of informed consent.

Investigators hypothesize that as informed consents have become more lengthy and complicated, in part due to required regulatory language and legal clauses inserted to protect the institution performing research, patient comprehension of the basic elements of informed consent has been hindered.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age
* Patients are receiving active treatment on an oncology clinical trial that utilizes chemotherapy, radiation, targeted agents, biologic therapy or hormonal therapy
* Patients must have been consented in English to an oncology treatment clinical study

Exclusion Criteria:

* Not meeting all eligibility criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer clinic
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2012-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Understanding of all elements of informed consent via questionnaire | 1 month
  Comprehension of the important elements of the informed consent forms using questionnaire

SECONDARY OUTCOMES:
Patient comprehension | every 6 months, up to 1 year
  Effectors of patient comprehension using questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Schumacher, Principal Investigator — Brown University
Locations (2):
- United States (2):
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island

REFERENCES:
- [Derived] Schumacher A, Sikov WM, Quesenberry MI, Safran H, Khurshid H, Mitchell KM, Olszewski AJ. Informed consent in oncology clinical trials: A Brown University Oncology Research Group prospective cross-sectional pilot study. PLoS One. 2017 Feb 24;12(2):e0172957. doi: 10.1371/journal.pone.0172957. eCollection 2017. PMID 28235011